CLINICAL TRIAL: NCT06650813
Title: Adapting the FACETS Fatigue Management Program to Sickle Cell Disease
Brief Title: Adapting the FACETS Program to Sickle Cell Disease
Acronym: Drépa-FACETS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Versailles Hospital (Other)
Collaborators: University Hospital, Grenoble (Other); University Grenoble Alps (Other); Paris Nanterre University (Other)
Responsible Party: Principal Investigator, Michalina DANNOUNE, Investigator Coordonnator, Versailles Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: P23/09 - Drépa-FACETS
Record Dates: First submitted 2024-10-15; First posted 2024-10-21 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Fatigue Symptom; Sickle Cell Disease
MeSH Terms: conditions — Fatigue; Anemia, Sickle Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with sickle cell disease (Experimental)
  Interventions: Other: Drépa-FACETS Program

INTERVENTIONS:
Other: Drépa-FACETS Program — Drépa-FACETS Program for Sickle Cell Disease

SUMMARY:
Adaptation of a fatigue management program combining the principles of cognitive-behavioral therapy and energy conservation strategies (FACETS program) for a population of adult patients with sickle cell disease (Drépa-FACETS program).

ELIGIBILITY:
Inclusion Criteria:

* Participant having freely given his oral agreement.
* Participant with a major sickle cell syndrome, regardless of genotype (e.g. SS, SC, Sbeta).
* Participant with a sufficient command of spoken and written French to take the assessments, complete the questionnaires, follow the program sessions and carry out the home exercises.

Exclusion Criteria:

* Participant with one or more severe psychiatric pathologies (e.g. severe depression, psychosis) that could interfere with the conduct of the study, in particular the primary and secondary endpoints.
* Participants with another chronic pathology causing fatigue.
* Participants in vaso-occlusive crisis (VOC) or hospitalization.
* Participant under legal protection (guardianship, curatorship, safeguard of justice, deprived of liberty).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2026-05-02 (Estimated); Study Completion 2026-05-02 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the FACETS program for adult sickle-cell patients | From the enrollment to the end of the protocol visits (10 weeks)
  Main criterion is assessing feasibility. Composite criterion including three sub-criteria are :
  1. Participation rate in the main sessions of the program. This criterion will be met if the participant attends at least 4 of the 6 sessions of the program.
  2. Success rate in completing home exercises. This criterion will be met if the participant completes at least 50% of the home exercises assigned at the end of each session.
  3. Acquisition of fatigue management skills. This criterion will be met if the participant has been able to implement one of the fatigue management techniques proposed by the Drépa-FACETS program in their daily life. The main criterion for evaluating the feasibility/acceptability of the DrépaFACETS program will be met if 2 of the 3 sub-criteria are met.

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Claire GAY, Pr, Study Director — Paris Nanterre University
Locations (2):
- France (2):
  - CHU Grenoble Alpes, Grenoble
  - Hospital Versailles, Le Chesnay